CLINICAL TRIAL: NCT00560040
Title: Myocardial Injury is Not Related to Training Levels Among Recreational Participants in the Silicon Valley Marathon
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Abbott Point of Care (Industry)
Other Study IDs: Miller 01
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-05

CONDITIONS: Troponin; Natriuretic Peptide, Brain; Exercise; Echocardiography
Keywords: Troponin; Natriuretic Peptide, Brain; Exercise; Echocardiography
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To determine if pre-race training effects heart damage induced by marathon running.

DETAILED DESCRIPTION:
Investigations have shown increases in cardiac markers consistent with myocardial injury and left ventricular dysfunction in both recreational and elite athletes after endurance exercise. Pre-race training is an important component of endurance events, yet its effect on cardiovascular injury is unclear. The present study aimed to evaluate the correlation between myocardial injury and training level in recreational marathon runners utilizing both objective and subjective measures.

ELIGIBILITY:
Inclusion Criteria:

* Any healthy male or female aged 18-65 planning to run the 2006 Silicon Valley Marathon.

Exclusion Criteria:

* Hypertension
* Hyperlipidemia
* Diabetes
* History of myocardial infarction or acute coronary syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-01; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne M Miller, MD, Principal Investigator — Stanford Hospital and Clinics